CLINICAL TRIAL: NCT01172379
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study of the Safety, Tolerability and Efficacy of E2007 in Parkinson's Disease Patients With "Wearing Off" Motor Fluctuations and "On" Period Dyskinesias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Eisai Medical Services, Eisai Inc
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-E044-204
Record Dates: First submitted 2010-07-26; First posted 2010-07-29 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental 1 (Experimental)
  Interventions: Drug: E2007
- Experimental 2 (Experimental)
  Interventions: Drug: E2007
- Experimental 3 (Experimental)
  Interventions: Drug: E2007
- Placebo Comparator (Placebo Comparator)
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: E2007 — Experimental 1 Drug: E2007
  0.5 mg 1 tablet per day
  Arms: Experimental 1
Drug: E2007 — Experimental 2 Drug: E2007
  1.0 mg 1 tablet per day
  Arms: Experimental 2
Drug: E2007 — Drug: E2007
  2.0 mg 1 tablet per day
  Arms: Experimental 3
Other: Placebo Comparator — Placebo 1 tablet per day
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and efficacy of E2007 in Parkinson's Disease patients who have "wearing off" motor fluctuations and "on" period dyskenisias.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, dose-ranging multicentre study with parallel groups. Patients will be equally randomized to receive 0.5 mg, 1 mg or 2 mg of E2007 or matching placebo for 12 weeks (84 days) in addition to their stable antiparkinsonian treatment. The study will involve two overnight in-patient stays. The first of these will be for 2 nights and 3 days and the second will be for 1 night and 2 days. The remainder of the study will be conducted on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with idiopathic PD fulfilling the Queen Square Brain Bank diagnostic criteria, with good response to levodopa.
2. Patients must be aged 30-75 inclusive. Patients aged between 76-80 (inclusive) may be enrolled with the prior agreement of the Study Medical Monitor.
3. Patients must have motor fluctuations of the wearing "off" type with the presence of at least two and half hours of "off" time during the waking day and at least 90 minutes of "off" time during the eight hour period following the morning dose of levodopa each per day as evidenced by history at Screening and confirmed by diary data collected between Screening and Baseline.
4. Patients must have clinically relevant dyskinesias during the "on" period following each morning dose of his/her current medication.
5. Patients must rate between II-IV on the Hoehn and Yahr scale when in an "off" state.
6. Patients must be taking levodopa at least three times daily.
7. Patients must have been on a fixed dose of any treatments for PD for at least 4 weeks prior to the Baseline Visit.
8. In the Investigator's opinion patients must be able to distinguish their own motor states and the absence or presence of dyskinesias.
9. Patients must be capable of giving full written informed consent.
10. In the Investigator's opinion patients must be of capable of completing patient diary cards according to instructions.
11. In the Investigator's opinion patients who are good candidates and able to complete the study.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Women of child-bearing potential unless infertile (including surgically sterile) or practicing effective contraception (e.g., abstinence, IUD or barrier method plus hormonal method). These patients must have a negative serum B-HCG test at the Initial Screening Visit and a negative urine pregnancy test at the Baseline Visit. These patients must also be willing to remain on their current form of contraception for the duration of the study. Postmenopausal women may be recruited but must be amenorrhoeic for at least 1 year to be considered of non-child bearing potential.
3. Fertile men not willing to use reliable contraception and fertile men with partners not willing to use reliable contraception.
4. Patients with a past or present history of drug or alcohol abuse.
5. Patients with a past (within one year) or present history of psychotic symptoms requiring antipsychotic treatment. Patients may be taking anti-depressant medication, however, the dose must be stable for 8 weeks prior to the Baseline Visit.
6. Patients with unstable abnormalities of the hepatic, renal, cardiovascular, respiratory, gastrointestinal, haematological, endocrine or metabolic systems which might complicate assessment of the tolerability of the study medication.
7. Patients with significantly elevated liver enzymes (abnormal bilirubin or seum transaminase levels of more than 1.5 times the upper normal limit).
8. Patients currently receiving treatment with medication that could significantly interfere with gastric absorption.
9. Patients with current or prior treatment (within 4 weeks prior to the Baseline Visit) with medication known to induce the enzyme cytochrome P450 3A4 including but not limited to: carbamazepine; dexamethasone; ethosuximide; phenobarbital; phenytoin; primidone; rifabutin; rifampacin; and St. John's Wort.
10. Current or prior treatment (within 4 weeks prior to Baseline Visit) with methyldopa, budipine, reserpine or intermittent use of liquid forms of levodopa or apomorphine.
11. Patients with previous stereotactic surgery (e.g., pallidotomy) for Parkinson's disease.
12. Patients receiving deep brain stimulation.
13. Patients who have received an investigational product within 12 weeks prior to Baseline Visit or patients that have participated in a previous study with E2007.
14. Patients with clinically significant cognitive impairment (MMSE ; 24 and/or fulfilling DSM IV criteria for dementia due to Parkinson's disease).
15. Patients with conditions affecting the peripheral or central sensory system unless related to Parkinson's disease (mild sensory or pain syndromes limited to off periods) that could interfere with the evaluation of any such symptoms caused by the study drug.
16. Patients with any condition that would make the patient, in the opinion of the Investigator, unsuitable for the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2
Dates: Start 2004-05; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Efficacy assessments: Parkinsonian symptomology will be recorded on an out-patient basis using patient diary cards (indicating "on" and "off" periods, sleep and dyskinesias). | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Webster, Study Director — Eisai Limited
Locations (33):
- Czechia (5):
  - Clinic of Neurology, Faculty Hospital Olomouc, Olomouc
  - Private Neurology Practise, Ostrava
  - Department of Neurology, Regional Hospital Pardubice, Pardubice
  - First Faculty of Medicine Charles University, Prague
  - Dept. of Neurology - Second Faculty of Medicine Charles University, Prague
- Centre D'Investigation Clinique Pavillon Riser - Hopital Purpan, Toulouse, France
- Germany (15):
  - Parkinson's Competence Network Germany Dept. of Neurology - Philipps-University Marburg, Marburg, Hesse
  - Humboldt Universit?t Charite Neurologische Klinik, Berlin
  - Klinikum der Friedrich-Wilhelms- Univerit?t Bonn, Bonn
  - Zentralkrankenhaus Reinkenheide Neurologische Klinik, Bremerhaven
  - Klinikum der Heinrich-Heine- Universit?t, D?sseldorf
  - Praxis, Erbach im Odenwald
  - Klinikum der Georg-August- Universit?t, G?ttingen
  - Universit?tskrankenh aus Hamburg Eppendorf, Hamburg
  - Krankenhaus Hanau, Hanau
  - Medizinische Hochschule Hannover, Hanover
  - Universit?tsklinikum Heidelberg, Heidelberg
  - Universit?tsklinikum, Homburg/Saar
  - Paracelsus-Elena-Kli nik, Kassel
  - Hopital Roger Salengro, Lille
  - Universit?tsklinikum Rostock Klinik f?r Neurologie, Rostock
- Italy (5):
  - Reparto di Neurologia - Ospedale Misericordia, Grosseto
  - Universit? di Napoli Federico II, Napoli
  - Unit? Operativa Parkinson e Disordini del Movimento, Pavia
  - Istituto Neuromed SRL Neurologia, Pozzilli
  - III Clinica Neurologica, Roma
- Serbia (3):
  - Militzary Medical Academy, Belgrade
  - Clinic of Neurology, Belgrade
  - Institute of Neurology, Belrade
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Mutua de Terrassa, Terrassa